CLINICAL TRIAL: NCT00498589
Title: A Controlled, Randomized, Double-blind, Multicenter Study, Comparing Methotrexate vs Placebo in Corticosteroid-dependent Ulcerative Colitis
Brief Title: Comparison of Methotrexate vs Placebo in Corticosteroid-dependent Ulcerative Colitis
Acronym: METEOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Franck Carbonnel, PU-PH, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GETAID 2006-1
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Methotrexate IM or SC 25 mg/week vs placebo IM or SC for 24 weeks
  Interventions: Drug: methotrexate
- 2 (Placebo Comparator): 1 IM or SC of placebo per week during 24 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methotrexate — 25 mg per week IM or SC during 24 weeks
  Arms: 1
Drug: placebo — one intramuscular injection per week
  Arms: 2

SUMMARY:
* PHASE: II
* TYPE OF STUDY : With direct benefit
* DESCRIPTIVE: Multicenter, randomized, double-blind study
* INCLUSION CRITERIA: Steroid-dependent ulcerative colitis
* OBJECTIVES: To show superiority of methotrexate vs placebo in inducing steroid-free remission in steroid-dependent ulcerative colitis
* STUDY TREATMENTS: Methotrexate 1 intramuscular injection (25 mg) per week Placebo 1 intramuscular injection per week
* NUMBERS OF PATIENTS: 55 patients in each group, i.e. a total of 110 patients
* INCLUSION PERIOD: 24 months
* STUDY DURATION: 36 months
* EVALUATION CRITERIA: Remission without steroids, immunosuppressives and without colectomy at 16 weeks of treatment.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease that slightly reduces life expectancy, strongly reduces its quality and can lead to serious complications such as acute colitis, dysplasia and colon cancer. About 40'000 patients are affected in France Among them, 15% suffer from a chronic active form that often leads to an extended steroid therapy, and its known side effects. Azathioprine has already proven its efficacy in this indication but brings a lasting remission without steroid in only 41% of the patients (1-4). What are the medications available for the patients who failed in maintaining a remission with azathioprine ? Cyclosporin is designed for severe or steroid-resistant forms. (5). The results of two recent studies have showed that infliximab is more efficacious than placebo in active UC (6, 7). Infliximab is expensive, its efficacy in steroid-dependent UC has not been specifically tested yet, and its tolerance on the long term remains uncertain. Methotrexate proved its efficacy in Crohn's disease with an intramuscular dose of 25mg/week (8). In UC a controlled trial has been negative with an oral dose of 12.5mg/week (9). Another study compared mercaptopurine, methotrexate (15mg/week) and 5-aminosalicylate in 72 steroid-dependent patients with CD or UC (10). The remission rates obtained were 58% after 30 weeks with methotrexate (not significantly different from 5-ASA) and 14% after 106 weeks (not significantly different from 5-ASA). Few data are available on the efficacy of methotrexate in UC, at a dose which is active in Crohn's disease (25mg intramuscular/week). Several uncontrolled series have been published, including 91 patients whose remission failed under azathioprine.

Methotrexate is cheap and its patent has fallen in the public domain. Only institutional research will be able to finance a study in this new indication.

This is a prospective, controlled, randomized, double-blind study of methotrexate with an intramuscular dose of 25mg/week vs placebo in patients with steroid-dependent UC.

This multicenter study will take place under the aegis of the Therapeutic Study Group for Inflammatory Digestive Diseases (G.E.T.A.I.D.) and with the help of the gastroenterologists network of the CIC. The issue of this study is important. If the hypothesis is borne out, a cheap, efficacious medication will be available for chronic active UC.

ELIGIBILITY:
Inclusion Criteria:

* UC diagnosed according to the Lennard-Jones criteria (Appendix 1) with endoscopic colorectal lesions, whatever their extension may be
* A Mayo Disease Activity Index £ 4, with no item >1 for the clinical part of the score and from 0 to 2 for the endoscopic part at the time of inclusion
* Steroid-dependence defined by at least 1 unsuccessful attempt to stop systemic steroid therapy during the last 12 weeks. Steroid therapy might have been completely stopped if it has been restarted within the last 30 days
* To be receiving a treatment of prednisone at a dose between 10 and 40mg, stable for at least 2 weeks at the time of inclusion
* Under an adequate contraception for male or female subjects of childbearing potential

Exclusion Criteria:

* Indication to a colectomy.
* Alcoholism (more than 21 glasses per week for male subjects and 14 glasses per week for female subjects). 1 glass corresponds to 3 cl of strong alcohol, 10 cl glass of wine or a half pint of beer.
* Pregnant or breast-feeding female subjects.
* No efficacious contraception.
* NSAIDS or cotrimoxazole intake upon inclusion, or probenecid intake within 1 month prior to inclusion.
* Anti-TNFa treatment within 2 months prior to inclusion.
* Azathioprine, mercaptopurine, cyclosporin or thalidomide within 1 month prior to inclusion.
* Modification of mesalazine or olsalazine dosage within 1 month prior to inclusion.
* Chronic (broncho) pneumopathy.
* Renal failure (creatinaemia > upper limit of normal laboratory values limit).
* Liver disease apart from primary sclerosing cholangitis.
* Unexplained rise higher than twice the normal level for transaminases, alkaline phosphatases and/or bilirubin.
* Folate level < normal level.
* Past history of malignant condition (including leukaemia, lymphoma and myelodysplasia) except for baso-cellular cutaneous cancers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-09; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Remission without steroids, immunosuppressives and without colectomy | week 16

CONTACTS AND LOCATIONS:
Overall Officials: Franck Carbonnel, Principal Investigator — CHU Besançon
Locations (22):
- University Hospital of Vienna, Vienna, Austria
- ULB - Cliniques Saint Luc, Brussels, Belgium
- France (16):
  - CHU Amiens - Hôpital Nord, Amiens
  - CH Avignon, Avignon
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - CHU Clermont-Ferrand - Hôpital Hotel Dieu, Clermont-Ferrand
  - APHP - Hôpital Beaujon, Clichy
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille - Hôpital Huriez, Lille
  - CHU Nantes - Hôpital Hôtel Dieu, Nantes
  - CHU Nice - Hôpital de l'Archet 2, Nice
  - APHP - Hôpital Saint Louis, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - APHP - Hôpital Cochin, Paris
  - CHU Bordeaux - Hôpital Haut L'Eveque, Pessac
  - CHU Rouen - Hôpital Charles Nicolle, Rouen
  - CHU St Etienne - Hôpital NOrd, Saint-Priest
  - CHU Toulouse - Hôpital Rangueil, Toulouse
- Sheba Medical Center, Tel Aviv, Israel
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano , Milano
  - Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo
- LUMC, Leiden, Netherlands

REFERENCES:
- [Derived] Carbonnel F, Colombel JF, Filippi J, Katsanos KH, Peyrin-Biroulet L, Allez M, Nachury M, Novacek G, Danese S, Abitbol V, Bossa F, Moreau J, Bommelaer G, Bourreille A, Fumery M, Roblin X, Reinisch W, Bouhnik Y, Brixi H, Seksik P, Malamut G, Farkkila M, Coulibaly B, Dewit O, Louis E, Deplanque D, Michetti P, Sarter H, Laharie D; European Crohn's and Colitis Organisation; Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives. Methotrexate Is Not Superior to Placebo for Inducing Steroid-Free Remission, but Induces Steroid-Free Clinical Remission in a Larger Proportion of Patients With Ulcerative Colitis. Gastroenterology. 2016 Feb;150(2):380-8.e4. doi: 10.1053/j.gastro.2015.10.050. Epub 2015 Nov 26. PMID 26632520